CLINICAL TRIAL: NCT01281059
Title: Prediction of Severity of Liver Disease Non Alcoholic Fatty Liver Disease in Patients With Suspected NAFLD by a 13C Octanoate Breath Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Meridian Bioscience, Inc. (Industry)
Responsible Party: Gadi Lalazar, Hadassah Medical Organization
Other Study IDs: 0429-10-HMO-CTIL
Record Dates: First submitted 2011-01-10; First posted 2011-01-21 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2011-08

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BreathID - Breath Test - 13C Octanoate

SUMMARY:
The Exalenz clinical investigation is a multicenter, non-randomized, blinded, study of the ¹³C-Octanaote breath test (OBT). The OBT is a non-invasive test for evaluation of disease severity in patients with suspected non alcoholic fatty liver disease (NAFLD) The purpose of the study is to demonstrate that the ¹³C-Octanaote Breath Test (OBT) can be used as an aid, in conjunction with other clinical information and medical history, for evaluating disease severity and detecting non alcoholic steatohepatitis(NASH) with a high probability.

Retrospective analysis based on multivariable analysis will determined if and which demographic, clinical and biochemical or imaging techniques data can assist in addition to the data derived from OBT in differentiation of NASH, NAFL and possibly normals.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (>18 years of age)
* Liver -biopsy ( at least 1.7 cm and 4 portal tracts) performed within 6 months of breath test or planned within the next 6 weeks, providing no treatment for liver disease was given between the biopsy and the OBT Any elevation of liver enzymes above the upper limit of normal (any or all of the following: AST,ALT, GGT, Alkaline phosphatase)
* At least one of the features of the metabolic syndrome

  * waist circumference > 100 cm for men, 88 cm for women
  * triglycerides > 150 mg/dl
  * fasting blood sugar > 110 mg/dl
  * HDL cholesterol < 40 mg/dl
  * blood pressure > 130/85 mm Hg
* No other known co-existent liver disease, excluded by appropriate serologic testing

Exclusion Criteria:

* Positive studies for any of the following:
* hepatitis C (PCR)
* hepatitis B (surface antigen or DNA)
* iron saturation > 60% + gene test for hereditary hemochromatosis
* antinuclear antibody at a titer > 1: 160 along with hypergammaglobulinemia and ALT levels>250 U/L

  * Patient has Alpha-1-antitrypsin level below lower limit of normal (< 150 mg/dl)
  * Patient has alcohol consumption > 20 gm/day for women and > 30 gm/day for men
  * Patient is pregnant
  * Patient has been taking known hepatotoxic drugs e.g. (e.g.acebutolol, indomethacin,phenylbutazone,allopurinol,isoniazid,phenytoin,atenolol,ketoconazole,piroxicam,carbamazepine,labetalol,probenecid,cimetidine,maprotiline,pyrazinamide,dantrolene, metoprolol,quinidine,diclofenac, mianserin)• Patients that have had more than 10% reduction in body weight since biopsy
  * Patient with known severe congestive heart failure (LVEF on echocardiogram < 20%)
  * Patient with known severe pulmonary hypertension (By echocardiogram, PAS >45 mmHg)
  * Patient with uncontrolled diabetes mellitus (HA1c>10)
  * Patient with previous surgical bypass surgery
  * Patient with extensive short bowel syndrome(>100 cm)
  * Patient currently receiving total parenteral nutrition
  * Patient is a recipients of any organ transplant
  * Patients that received any anti-viral treatment or any other liver therapy between the time of the biopsy and the breath test.
  * Women who are pregnant
  * Patients with an acute current exacerbation of chronic obstructive pulmonary disease or bronchial asthma.
  * Patient has taken drugs that can interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine.
  * Patients unable or refuse to sign informed consent
  * Patients that based on the opinion of the investigator should not be enrolled into this study
  * Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel